CLINICAL TRIAL: NCT00602212
Title: The Potential of Virtual Reality as Anxiety Management Tool: a Randomised Controlled Study in a Sample of Patients Affected by Generalized Anxiety Disorder
Brief Title: Virtual Reality as Anxiety Management Tool for Generalized Anxiety Disorder
Acronym: INTREPID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03E701; IST-2002-507464 (Other Grant/Funding Number: European Union - IST Programme - FP5)
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Last update posted 2011-09-09 (Estimated); Status verified 2008-01

CONDITIONS: Generalized Anxiety Disorder
Keywords: generalized anxiety disorder (GAD)
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Biofeedback, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VR + Mobile Phone without Biofeedback (Active Comparator): In this experimental condition patients received an eight-session VR-based treatment including relaxation and exposure
  Interventions: Behavioral: relaxation with virtual reality (VR); Behavioral: relaxation and biofeedback virtual reality
- VR + Mobile Phone with biofeedback (Experimental): The patients experienced the same protocol described above, but with the biofeedback support. Specifically, in the sessions with the therapist, HR variations were used to modify specific features of the virtual environment:
  Interventions: Behavioral: relaxation with virtual reality (VR); Behavioral: relaxation and biofeedback virtual reality

INTERVENTIONS:
Behavioral: relaxation with virtual reality (VR) — VR relaxing environment and audio-visual mobile narratives will be used to teach patients how to relax themselves
  Other Names: relaxation; virtual reality
Behavioral: relaxation and biofeedback virtual reality — The patients experienced the same protocol described above, but with the biofeedback support. Specifically, in the sessions with the therapist, HR variations were used to modify specific features of the virtual environment:
  Other Names: relaxation; virtual reality; biofeedback

SUMMARY:
Generalized Anxiety Disorder (GAD) is a psychiatric disease characterized by long-lasting anxiety that is not focused on a specific object or situation. According to the DSM-IV-TR the essential feature of GAD is at least six months of "excessive anxiety and worry" about a variety of events and situations. Anxiety and worry are often accompanied by a variety of physical symptoms like restlessness, being easily fatigued, difficulty concentrating, irritability, muscle tension and disturbed sleep. The high prevalence of GAD in the general population and the severe limitations it causes point out the necessity to find new strategies to treat it in a more efficient way. Within the treatment of GAD, physical (relaxation and controlled breathing), behavioral (visualization and controlled exposure) and cognitive control strategies (challenging negative thoughts) represent a key part of the treatment, even if they are hard to be learned. Given the features of this disease and its pervasive effect on patient's personal, occupational and affective life, we thought it could benefit from an ubiquitous treatment.We suggested, then, to improve the treatment of GAD through the use of a biofeedback enhanced virtual reality (VR) system used for relaxation, controlled exposure and SIT. The use of SIT in the context of GAD is motivated by the acknowledgment that sometimes stressors can't be avoided or altered and then patients can't apply strategies focused on finding solutions. In these instances, coping effort should be directed to emotionally palliative set of responses such as acceptance, reframing and perspective thinking. All these cognitive changes are facilitated if a concomitant relaxation is induced. The treatment involves two virtual reality components:

I) an immersive virtual reality system experienced in the therapist's office;

II) a mobile exposure system allowing patients to perform the virtual experience in an outpatient setting. The role of the mobile exposure system is the following:

* To present and structure emotionally relevant contents in an ubiquitous context.
* To verify the compliance of the patient and eventually alert patient/therapist;
* To track in real-time the emotional level of the patient and record it for later assessment by the therapist;
* To provide a feedback to the patient able to help him in coping with the contents;
* To automatically contact the therapist if the emotional level is higher than a preset cut-off value defined by the therapist.

DETAILED DESCRIPTION:
The patients were randomly assigned to the following groups: (1) the VR and Mobile group (VRMB) including biofeedback - 7 subjects; (2) the VR and Mobile group (VRM) without biofeedback - 9 subjects; (3) the waiting list (WL) group - 8 subjects:

1. Virtual Reality + Mobile Phone without Biofeedback Condition (VRM). In this experimental condition patients received an eight-session VR-based treatment including relaxation and exposure. In sessions 1 to 6, the patient explored a beautiful VR tropical island (experienced with a head-mounted display and head-tracking) following a predefined path leading to different relaxing areas: Campfire, Beach and Waterfall. In these areas the patients started to relax by observing the flickering campfire, watching waves lapping gently on a shore, or looking to the waterfall and fish pond. Each experience was supported by an audio narrative based on progressive muscle relaxation and/or autogenic techniques. All the environments were developed by the ESIEA INTREPID team (J.L. Dautin, J. Ardouin, F. Crison and M. Le Renard -www.esiea.fr) using the 3DVIA 4.1 Virtools toolkit by Dassault Systèmes - www.virtools.com.To improve the efficacy of the training and to increase the effects of relaxation, patients experienced at home, using a mobile phone, on a non-navigable version of the same virtual reality environment experienced during the therapy. The patient was asked to train relaxation abilities at least once a day for the entire duration of the treatment following the treatment plan provided by the therapist. In session 7 and 8 the patients explored again the island reaching a Gazebo in which they are exposed to pre-selected words or images related to their personal stressful events. The patients were then asked to use the learned relaxation techniques to cope with them.
2. Virtual Reality + Mobile Phone with Biofeedback Condition (VRMB). The patients experienced the same protocol described above, but with the biofeedback support (see Figure 2). Specifically, in the sessions with the therapist, HR variations were used to modify specific features of the virtual environment:

   1. Campfire (sessions 1-2). HR controls the fire intensity: a reduction of the patient's physiological activation reduces fire intensity until it disappears;
   2. Beach (sessions 3-4). HR controls the movement of the waves: a reduction of the patient's physiological activation reduces the movement of the waves until the ocean becomes completely calm;
   3. Waterfall (sessions 5-6): HR controls the movement of the water: a reduction of the patient's physiological activation reduces the movement of the water until the water flow becomes completely still;
   4. Gazebo (sessions 7-8): HR controls the size of a stressful image or video: a reduction of the patient's physiological activation reduces the size of the stimulus until it disappears. This exercise is designed following the procedure of SIT.
3. Waiting List Condition (WL). This was a control condition, in which patients were included in a waiting list and not received any kind of relaxation training.

ELIGIBILITY:
Inclusion Criteria:

1. Primary diagnosis of GAD
2. Requesting treatment for their GAD
3. Older than 17 and younger than 70; (4) no change in dose of psychotropic medications 1 month before inclusion

Exclusion Criteria:

1. Depressive disorder preceding the current episode of GAD or requiring immediate treatment
2. Behavior therapy received for their GAD
3. Evidence of organic mental disorders accounting for the complaints, mental retardation, psychotic disorders, alcohol or drug dependence
4. Migraine, headache, seizure disorder, and vestibular abnormalities since they represent significant contraindications for the use of VR.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-02; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
level of anxiety measured by: psychometric questionnaires (PSWQ, BAI, Anti, CID, STAI) and psychophysiological measures ((skin conductance response (SCR), muscle tension, heart and respiratory rates) | immediately before and after each treatment session. At follow up (6 and 12 months)

SECONDARY OUTCOMES:
subjective measures (diary) | during the treatment and during the follow up period

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Riva, Phd, Study Director — Istituto Auxologico Italiano; Alessandra Gorini, PsyD, Principal Investigator — Istituto Auxologico Italiano
Locations (1):
- Istituto Auxologico Italiano, Milan, Italy

REFERENCES:
- [Background] Riva G, Gorini A, Gaggioli A. The Intrepid project - biosensor-enhanced virtual therapy for the treatment of generalized anxiety disorders. Stud Health Technol Inform. 2009;142:271-6. PMID 19377166
- [Background] Gorini A, Riva G. The potential of virtual reality as anxiety management tool: a randomized controlled study in a sample of patients affected by generalized anxiety disorder. Trials. 2008 May 5;9:25. doi: 10.1186/1745-6215-9-25. PMID 18457580
- [Result] Repetto C, Gorini A, Vigna C, Algeri D, Pallavicini F, Riva G. The use of biofeedback in clinical virtual reality: the INTREPID project. J Vis Exp. 2009 Nov 12;(33):1554. doi: 10.3791/1554. PMID 19915521
- [Result] Repetto C, Gorini A, Algeri D, Vigna C, Gaggioli A, Riva G. The use of biofeedback in clinical virtual reality: the intrepid project. Stud Health Technol Inform. 2009;144:128-32. PMID 19592748
- [Derived] Gorini A, Pallavicini F, Algeri D, Repetto C, Gaggioli A, Riva G. Virtual reality in the treatment of generalized anxiety disorders. Stud Health Technol Inform. 2010;154:39-43. PMID 20543266